CLINICAL TRIAL: NCT06085040
Title: Adaptations métaboliques, énergétiques et Nutritionnelles à la Perte de Poids Chez l'Adolescent Avec obésité : rôle du degré de Perte de Poids. Etude POWELL-2
Brief Title: Pedicatric Obesity - Weight - Energy - Loss - Load
Acronym: POWELL-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2023 BOIRIE 2
Record Dates: First submitted 2023-10-11; First posted 2023-10-16 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: Multidisciplinary weight loss

INTERVENTIONS:
Behavioral: Multidisciplinary weight loss — 12-months multidisciplinary behavioral intervention combining physical activity (3 times 60 minutes per week), nutritional guidance (balanced meals) and psychological support (60 minutes per week)

SUMMARY:
Although multidisciplinary treatment of pediatric obesity has shown its effectiveness in leading to weight loss and improvement in the physical, mental and social health of children and adolescents; maintaining these benefits remains a real challenge. Indeed, the literature clearly shows a short- to medium-term increase in weight, the mechanisms of which have yet to be identified in order to prevent it. Although cognitive, behavioral and nutritional adaptations have been highlighted to explain this weight regain, metabolic and energetic adaptations also seem to contribute. Indeed, a reduction in resting and total energy expenditure has been shown (in connection with changes in body composition and in particular lean mass), but also of the energy cost during locomotion and mobility, thus altering the daily energy balance. These energy adaptations are also accompanied by a modification in the use of energy substrates due to a modification of muscular metabolic flexibility in particular, leading to a reduction in lipid oxidation in favor of carbohydrates. Importantly, if this reduction in the use of lipids generates a counterproductive sparing of adipose tissue, thus slowing down weight loss, the increase in carbohydrate oxidation leads to an intensification of orexigenic signals at the central level, promoting nutritional compensations and positive energy balance and therefore contributing to weight regain.

Thus, these adaptations of energy metabolism and their interactions with dietary control seem to be at the heart of the mechanisms limiting the success of obesity treatment, favoring weight gain. If these observations were made at the end of treatment programs lasting several weeks to months, a recent clinical work highlights the need to consider the kinetics and temporality of weight loss (weight loss variability and rate of weight loss), so as to identify the crucial stages where these adaptations take place and thus prevent their energy consequences.

Thus, the main objective of this project is to study total energy adaptations (energy and nutritional metabolism) at rest but also during locomotion, during the central phase of weight loss of adolescents with obesity, as well as during phases of weight regain. Ultimately, the objective of this study is to better understand energetic adaptations to weight loss and the implication of the degree of weight loss in order to study the role of the interaction between these adaptations and the degree of weight loss on the success of programs and on the profiles of "weight maintainers" or "weight regainers".

DETAILED DESCRIPTION:
After an inclusion visit to ensure the adolescents' ability to complete the entire study, they will then complete 6 experimental visits: i) before their weight loss program (T0); ii) then a visit after a weight loss of 5% (T-5%); iii) after losing 10% of their weight (T-10%); iv) after 12 weeks of treatment (T1); v) after 24 weeks of treatment (T2) and; vi) after 4 months of post-intervention follow-up (T3).

During each of these visits, densitometric (body composition and bone structure) and anthropometric (height, body mass, waist circumference, hip circumference) measurements will be taken. Their resting metabolism as well as their energy consumption during a low-intensity incremental walking exercise will be measured by indirect calorimetry. Their sleep metabolism will be assessed over one night using Dreem headbands and their dietary control assessed during a calibrated test meal (satiety quotients and food reward). Their perception of health and quality of life, as well as the perception of their physical condition and their dietary profiles will be evaluated by questionnaire. The cardiovascular profile will also be assessed by measuring sinus variability, hepatic steatosis, arterial stiffness and the resistance and reactance of the respiratory system. Finally, a fasting blood sample will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 12 to 16 years (maturation 3-5 according to Tanner stages), having a body mass index (BMI) greater than the 97th percentile according to national curves.
* Able to give informed consent (parental authorization and assent of the minor) to participate in the research.
* Person subject to a Social Security system

Exclusion Criteria:

* Medical or surgical history judged by the investigator to be incompatible with the study.
* Presence of diabetes, and any other pathology limiting the application of one or the other strategy being tested.
* Subjects currently undergoing energy restriction or a weight loss program through physical activity at the time of inclusion or during the last 6 months.
* Taking medications that may interfere with study results
* Subjects with cardiovascular problems, we are talking here about subjects with a history of cardiovascular and/or neurovascular pathology, as well as subjects presenting cardiovascular and/or neurovascular risk factors (excluding obesity/ overweight).
* Surgical intervention within the previous 3 months.
* Pregnant or breastfeeding adolescents
* Person under guardianship/curatorship or safeguard of justice
* Participant's refusal to participate
* Refusal of consent (parental authorization) from holders of parental authority
* Person in period of exclusion from another study
* Consumption of tobacco or alcohol.
* Parents under curatorship/tutorship or legal protection.
* Special diet.
* Participation in regular and intense physical and sporting activities for more than two hours per week.
* Refusal of participation by legal representatives.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2024-06-25 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Body Weight | Before weight loss ; after a 5 and 10 % weight loss, after 6 months of weight loss, after 12 months of weight loss, After a 4-month follow-up
  The adolescents weight will be assessed
Body composition | Before weight loss ; after a 5 and 10 % weight loss, after 6 months of weight loss, after 12 months of weight loss, After a 4-month follow-up
  Fat Mass and fat Free Mass by absorptiometry

SECONDARY OUTCOMES:
resting energy expenditure | Before weight loss ; after a 5 and 10 % weight loss, after 6 months of weight loss, after 12 months of weight loss, After a 4-month follow-up
  Energy expenditure during a 20-minute rest using an indirect calorimeter
Exercise energy expenditure | Before weight loss ; after a 5 and 10 % weight loss, after 6 months of weight loss, after 12 months of weight loss, After a 4-month follow-up
  Energy expenditure during a 20-minute walking exercise using an indirect calorimeter
Food reward | Before weight loss ; after a 5 and 10 % weight loss, after 6 months of weight loss, after 12 months of weight loss, After a 4-month follow-up
  Liking and wanting for food in the fasted state using a computerized task
cardiometabolic profile | Before weight loss ; after a 5 and 10 % weight loss, after 6 months of weight loss, after 12 months of weight loss, After a 4-month follow-up
  Classical fasting blood profile

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France